CLINICAL TRIAL: NCT01734252
Title: A Pilot Trial to Assess the Efficacy of Argatroban (Argatra®) in Critically Ill Patients With Heparin Resistance
Brief Title: Argatroban in Critically Ill Patients With Heparin Resistance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Dietmar Fries, M.D., Coordinating and Principal Investigator, Medical University Innsbruck
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ArgHeR
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Achievement of a Sufficient Thrombosis Prohpylaxis in Clitically Ill Patients With Heparin Resistance
MeSH Terms: interventions — argatroban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Treatment (No Intervention): If a Heparin resistance appears and the patient meets the inclusion and exclu-sion criteria, he/she will be enrolled. The Heparin administration will be contin-ued and, if necessary increased. Hereby the maximum heparin dose is 1.500 IU per hour.
- Treatment with Argatroban (Experimental): If a Heparin resistance appears and the patient meets the inclusion and exclu-sion criteria, he/she will be enrolled. The Heparin administration will be stopped and Argatroban will be given and adjusted until the target aPTT-range is achieved.
  Interventions: Drug: Argatroban

INTERVENTIONS:
Drug: Argatroban — Start: Argatroban dose is 0.05 µg/kg/min (patients with hepatic impairment, after cardiac surgery) until maximum: 10 µg/kg/min
  Arms: Treatment with Argatroban

SUMMARY:
Critically ill patients with high risk for thrombosis or tromboembolic events with the presence of heparin resistance, treated at the Department for General and Surgical Critical Care Medicine of the Medical University Innsbruck, Austria will be enrolled in the study when meeting the inclusion- and exclusion criteria. If a patient meets the inclusion criteria and is recruited for the study, the patient will be randomized either to Group A or Group H.

All patients have to achieve a prophylactic aPTT-target range of an aPTT-level of 45 - 60 sec (Pathromtin® SL) within 6 to 8 hours.

Randomisation Group A:

If a Heparin resistance appears and the patient meets the inclusion and exclu-sion criteria, he/she will be enrolled. The Heparin administration will be stopped and Argatroban will be given and adjusted until the target aPTT-range is achieved.

Randomisation Group H - Standard therapy:

If a Heparin resistance appears and the patient meets the inclusion and exclu-sion criteria, he/she will be enrolled. The Heparin administration will be contin-ued and, if necessary increased. Hereby the maximum heparin dose is 1.500 IU per hour.

Therapy failure Group H:

Primary target failure at Visit 3 (6-8 hours):

If a patient of Group H does not achieve the target-aPTT within 6-8 hours, he/she will switch to Group A and will start with T1 (Baseline) and will follow the visits according to Group A until the final Visit 9 (T1 / day 30).

Maintenance failure after Visit 3:

Maintenance failure after 6-8 hours is defined as non-maintenance of the tar-get-aPTT until day 7 with a max. heparin dosage of 1.500 IU per hour. In this case, heparin therapy has to be changed to Argatroban.

The patient will start with T1 (Baseline) and will follow the visits according to Group A until the final Visit 9 (day 30) counting from the Baseline of Group A.

Therapy failure Group A:

If a patient of Group A does not achieve the target-aPTT within 6-8 hours or cannot maintain the target-aPTT in spite of reaching the maximum dosage of 10µg/kg/min during the further study period, the patient automatically drops out of the study.

The same is effective for patients who switched to the Group A after a therapy failure in Group H.

General:

Two hours after starting the Baseline investigations, patient's parameters in-cluding blood collections will be measured for the second time (T2). Additional measurements will be made at 6-8 hours (T3), 24 hours (T4), 48 hours (T5), 5 days (T6) after start of study drug and on day 7 before (T7) stop of study medication and 6h (T8) after stop of study medication. 30 days after inclusion in the study, a final investigation is planned (T9).

ELIGIBILITY:
Inclusion Criteria:

* Patient at risk for thrombosis or thromboembolic complications with the need of prophylactic antithrombotic therapy
* Age: 18 - 85 years
* Prohylactic anticoagulation (aPTT: 45 - 60 sec) is not achieved with a heparin dosage of 1.200 IU per hour after two hours of infusion

Exclusion Criteria:

* If patient needs an aPTT-level > 60 sec for any reason
* Active bleeding
* Risk for bleeding higher than risk of thromboembolic event as anticipated by the physician
* Surgical procedure with the need for interruption of antithrombotic therapy within the next 24 hours
* Inevitable lethal course
* Severe Liver failure: Quick < 30 %
* Pregnancy
* Planned peridural or spinal anaesthesia during the study
* Patient with known refusal of a participation in this clinical trial
* Active participation in another clinical trial
* Any condition, including the presence of laboratory abnormalities, which would place the subject at unacceptable risk if he/she were to participate in the study or confound the ability to interpret data from the study
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-07-29 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2016-04-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who achieved the prophylactic aPTT-range within 6 - 8 hours (Visit 3). | The average period for the measurement (aPTT) of the primary outcome is 7 hours. Timepoints of measurements are at Baseline (hour 0) and after 6-8 hours.
  The primary measure is to achieve a prophylactic anticoagulation level within 7(+/-1) hours after Baseline. The parameter to define the anticoagulation level is aPTT and will be measured at 7(+/-1) hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Innsbruck / Department for General and Surgical Intensive Care Medicine, Innsbruck, Austria

REFERENCES:
- [Derived] Bachler M, Hell T, Bosch J, Treml B, Schenk B, Treichl B, Friesenecker B, Lorenz I, Stengg D, Hruby S, Wallner B, Oswald E, Strohle M, Niederwanger C, Irsara C, Fries D. A Prospective Pilot Trial to Assess the Efficacy of Argatroban (Argatra(R)) in Critically Ill Patients with Heparin Resistance. J Clin Med. 2020 Mar 31;9(4):963. doi: 10.3390/jcm9040963. PMID 32244368